CLINICAL TRIAL: NCT05585827
Title: A Decentralized Trial of Individual Video-assisted Cognitive Behavioural Therapy for Depressive Disorder in Parkinson's Disease.
Brief Title: Online Cognitive Behavioral Therapy for Depressive Symptoms in Parkinson's Disease
Acronym: ePark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 3414-3414
Record Dates: First submitted 2022-09-20; First posted 2022-10-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; Depressive Symptoms; Anxiety
Keywords: Parkinsons disease; Neuropsychiatry; Cognitive behavioral therapy
MeSH Terms: conditions — Parkinson Disease; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a online, randomized delayed start trial of the effectiveness of e-CBT for PD patients with depressive symptoms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate eCBT with concurrent TAU (Experimental): Those randomized into the this group will get immediate e-CBT with TAU.
  Interventions: Behavioral: Online cognitive behavioral therapy
- Delayed eCBT with concurrent TAU (No Intervention): Those randomized to the delayed arm of the study, will receive TAU and wait 14 weeks before receiving the intervention. TAU will include ongoing review by the patient's primary care physician, neurologist and PD nurse. TAU does not preclude clinically indicated adjustments to medication or specialist referrals but physicians are asked to keep medication constant if possible. For patients with PD ordinary treatment includes a multitude of interventions, including pharmacological treatment, speech therapy and physical therapy. Pharmacological interventions include the use of dopaminergic treatments, including levodopa and dopamine agonist use, with adjunct use of monoamine oxidase B-inhibitors.

INTERVENTIONS:
Behavioral: Online cognitive behavioral therapy — The e-CBT treatment manual is an adjusted version of a previously published treatment manuals for neuropsychiatric symptoms in PD, which is tailored to the preferences and needs for each participant. This manual encompass both modules from manuals for depression in PD and anxiety in PD. Individualization is ensures by including several interventions modules in the manual, wherein 5 sessions are considered "core modules", and four modules that can be offered depending on the patients individual needs. The participant may include partners or caregivers. The treatment is schedules to be completed within 13 weeks, with maximum ten sessions during this period. Following each e-CBT session, the participant will be asked to complete a short survey evaluating the acceptability and relevance of the session, and evaluate the therapeutic alliance.
  Arms: Immediate eCBT with concurrent TAU

SUMMARY:
More than 1 million people in Europe suffer from Parkinson's disease (PD), a brain disorder manifesting with a motor syndrome and several non-motor features. Neuropsychiatric symptoms, like anxiety and depression, are common in patients with PD, and has profound effects on quality of life and activities of daily living of the patient, and caregiver burden. Cognitive behavioral therapy (CBT) has proven efficient for depressive symptoms, but treatment availability to the general patient with PD is low. Thus, there is an urgent need for individualized remote approaches that can be of benefit to patients on a national scale. This study is a remote, randomized delayed start trial of the effectiveness of videoconference based cognitive behavioral therapy (eCBT) for PD patients with depressive symptoms. N=120 participants with PD and depressive symptoms will be recruited from neurological clinics across four health regions in Norway and self-reference, and randomized into two arms: (A) immediate eCBT with concurrent with TAU and (B) a delayed start (14 weeks) of eCBT with TAU alone. Patients will be assessed at baseline before allocation to treatment, with followed up evaluations 14, 28 and 42 weeks after baseline. The trial is designed as a state-of-the-art remote clinical trial, that can be easily implemented existing health services, resulting in a rapid implementation and improvement of treatment for patients with PD, and potentially large translational value to other brain disorders.

DETAILED DESCRIPTION:
We will conduct a remote, randomized controlled trial with delayed start, in order to:

1. Assess the 14-week effectiveness of eCBT for depressive symptoms for patients with PD.
2. Assess long-term outcomes, and predictors of long-term outcomes, of eCBT for depressive symptoms in PD.
3. Explore the impact and clinical correlates of working alliance in eCBT in patients with PD.

   For the first aim, we hypothesize that:

   i. 10 week eCBT will reduce the self-reported severity of depressive symptoms in patients with PD after 14 weeks, as compared to patients in a delayed start group, receiving treatment as usual (TAU).

   ii. 10 week eCBT will reduce the observed severity of depressive symptoms in patients with PD after 14 weeks, as compared to patients in a delayed start group, receiving TAU.

   i. 10 week eCBT will improve self-reported health related quality of life measured with The 8-item PD Questionnaire after 14 weeks, as compared to patient in a control group receiving TAU.

   For the second aim, we hypothesize:

   ii. Participants with 42 week follow up has lasting effects of eCBT, when compared to participants with 28 week follow up.

   iii. Long-term treatment response from eCBT for depressive symptoms, is predicted by the level of comorbid symptoms of anxiety and impulse control disorders at baseline.

   iv. Long-term treatment response from eCBT for depressive symptoms, is predicted by the level of comorbid symptoms of anxiety and impulse control disorders at the time of treatment completion.

   For the third aim, we hypothesize:

   i. The interrater agreement between patients and CBT therapist on working alliance will be a significant predictor of the acceptability of eCBT, as defined by patient reported experience measures.

ELIGIBILITY:
Inclusion Criteria:

* Signed written electronic consent;
* Confirmed PD clinical diagnosis based on self-report;
* A verified diagnosis of depression, according to previously published criteria;
* Age 35 to 85 years;
* Stable medication and mental health regiment (including antidepressants ≥ 6 weeks);
* Internet access from a computer or tablet.

Exclusion Criteria:

* Cognitive impairment as defined by Montreal Cognitive Assessment (MoCA) Blind version scores of <18;
* Suicidal thoughts with plan and intent (clinical interview);
* Medically unstable;
* Currently receiving psychotherapeutic treatment;
* History of bipolar or psychotic disorders;
* Does not speak Norwegian;
* A history with neurosurgery (like deep brain stimulation);
* No familiarity and/or access to a computer or tablet with camera, or internet access.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Change in The Clinical Global Impression scale (CGI) score | Baseline (BL) to 14 weeks
  A clinical-rated measure of general symptom severity of neuropsychiatric symptoms.
Change in the Hospital Anxiety and Depression Scale (HADS), score | Baseline (BL) to 14 weeks
  HADS is a commonly used self-report 14-item scale for the assessment of anxiety and depression in PD.
Change in the 8-item PD Questionnaire | Baseline (BL) to 14 weeks
  The 8-item version of the Parkinson's Disease Questionnaire (PDQ-8) is a shortened version of the 39-item Parkinson's Disease Questionnaire (PDQ-39). It was developed to reduce the respondent burden and increase convenience for use among persons with Parkinson's Disease in clinical settings.

SECONDARY OUTCOMES:
Change in the Automatic Thoughts Questionnaire-30- Negative (ATQ-30-N) score | Baseline, 14, 28 and 42 weeks
  is a 30-item self-report measure of the frequency of automatic negative thoughts associated with depression and anxiety.
Change in the The Behavioural Activation for Depression Scale (BADS) score | Baseline, 14, 28 and 42 weeks
  BADS is a 25-item self-report measure developed to measure the changes in activation and avoidance over the course of treatment of depression.
Change in The 39-item PD Questionnaire (PDQ-8) score | Baseline, 14, 28 and 42 weeks
  The PDQ-8 is a brief, valid and reliable patient reported outcome measure instrument to assess HRQoL in patients with PD with good concordant validity to generic HRQoL-scales.
The Negative Effects Questionnaire (NEQ) | 14, 28 and 42 weeks
  NEQ is a 20 item self-report questionnaire measuring adverse and unwanted effects for psychological treatments.
Change in the Parkinson Anxiety Scale (PAS) score | Baseline, 14, 28 and 42 weeks
  PAS is a 12-item self-report questionnaire measuring anxiety symptoms in patients with PD.
Patient reported experience measure (PREM): | 14, 28 and 42 weeks
  Participants experiences will be assessed with a six item questionnaire, scored on a visual analogue scale anchored with ''not at all'' to ''very much''. The questionnaire is comprised of six question indices: (1) interesting, (2) easy to understand, (3) useful, (4) extent to which the intervention provided novel information, (5) satisfaction, and (6) relevance.
Patient version of the Working Alliance Inventory (WAI): | 14, 28 and 42 weeks
  WAI is a 12-item questionnaire evaluating the working alliance between patients and the CBT-therapist.
Change in the Parkinson's Disease Impulsive-Compulsive Disorders Questionnaire Rating scale (QUIP-RS) score | Baseline, 14, 28 and 42 weeks
  QUIP-RS is a quick assessment of the severity of impulsive and compulsive behaviors in Parkinsons disease.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander H Erga, PhD, Principal Investigator — Norwegian Centre for Movement Disorders, Stavanger University Hospital
Locations (1):
- Stavanger University Hospital, Norwegian Centre for Movement Disorders, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erga AH, Alves G, Leentjens AFG. The ePark study protocol: A decentralized trial of individual video-assisted cognitive behavioural therapy for depressive disorder in Parkinson's disease. Contemp Clin Trials Commun. 2023 Feb 3;32:101080. doi: 10.1016/j.conctc.2023.101080. eCollection 2023 Apr. No abstract available. PMID 36817735
- [Background] Erga AH, Alves G, Leentjens AFG. Corrigendum to "The ePark study protocol: A decentralized trial of individual video-assisted cognitive behavioural therapy for depressive disorder in Parkinson's disease" [Contemp. Clinic. Trials Commun. 32 (2023) 101080]. Contemp Clin Trials Commun. 2023 Aug 29;35:101205. doi: 10.1016/j.conctc.2023.101205. eCollection 2023 Oct. PMID 37745287
- See also: Study website (Norwegian) — https://www.helse-stavanger.no/fag-og-forskning/kompetansetjenester/senter-for-bevegelsesforstyrrelser/epark-studien